CLINICAL TRIAL: NCT00553592
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel, Multicenter Study of the Safety and Efficacy of Two Dosages of Bicifadine SR in Adult Outpatients With Chronic Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Double Blind RCT of Bicifadine SR in Outpatients With Chronic Neuropathic Pain Associated With Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XTL Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XTL B07-001
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — bicifadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Drug (Experimental): Bicifadine
  Interventions: Drug: Bicifadine
- Drug: 2 (Experimental): Bicifadine
  Interventions: Drug: Bicifadine
- Control (Placebo Comparator): Placebo of Bicifadine
  Interventions: Drug: Bicifadine

INTERVENTIONS:
Drug: Bicifadine — 600mg/day
  Arms: Drug
Drug: Bicifadine — placebo tablet
  Arms: Control
Drug: Bicifadine — 1200 mg
  Arms: Drug: 2

SUMMARY:
To compare the efficacy of two dosages (600mg/day and 1200mg/day) of bicifadine SR with placebo for 14 weeks in reduction of chronic neuropathic patin (measured by a daily rating of pain intensity) associated with diabetic periperal neuropathy in adult outpatients.

To compare the tolerability of two dosages of bicifadine SR with placebo in adult outpaitens treated for chronic neuropathic pain for 14 weeks associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Diagnosis of type-1 or type 2 non-insulin dependent diabetes mellitus
* Chronic bilateral pain due to diabetic neuropathy
* Pain for at least six months
* Primary pain is located in the feet
* Others-contact site for information

Exclusion Criteria:

* Symptoms of other painful conditions
* Presence of amputations other than toes
* Clinically significant psychiatric or other neurological disorder
* Use of certain medications
* Clinically important other diseases
* Pregnancy
* History of alcohol or narcotic abuse within two years
* Others-contact site for information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2007-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pain and Safety | 14 weeks

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement, McGill Pain Questionnaire, Amount of Rescue Medication Used for Pain, Quality of Life Survey (SF-36), Patient Global Impression of Change | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Roffman, PhD, Study Director — XTL Bio
Locations (1):
- Four Rivers Clinical Research, Paducah, Kentucky, United States

REFERENCES:
- See also: Sponsor's website — http://www.xtlbio.com